CLINICAL TRIAL: NCT03592901
Title: Phantom Limb Experience After Brachial Plexus Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, Jack Tsao, MD, DPhil, University of Tennessee
Other Study IDs: 16-04696-XP
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Phantom Limb; Brachial Plexus Block
MeSH Terms: conditions — Phantom Limb | interventions — Brachial Plexus Block

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BPA Patients: Participants that are receiving brachial plexus anesthesia for a previously planned shoulder surgery.
  Interventions: Drug: brachial plexus anesthesia

INTERVENTIONS:
Drug: brachial plexus anesthesia — Anesthesia to some part of the brachial plexus prior to surgery. Patients are already receiving this regardless of participation in study.

SUMMARY:
This study examines the sensations felt by patients receiving brachial plexus anesthesia for shoulder surgeries.

DETAILED DESCRIPTION:
1. Purpose:

   The purpose of this study is to investigate whether phantom limb pain and/or sensations can arise after induction of BPA prior to upper extremity surgery. In addition, this study aims to investigate if there is cortical remapping of the hand sensation onto the face before and after surgery. The outcome of this research will provide insight into the characteristics of cortical reorganization and how this correlates to phantom limbs, phantom pain, and hand-to-face remapping.
2. Rationale, Research has yet to elucidate the etiology of phantom limb experiences, and the debate over peripheral or central nervous system mechanisms remains contentious. Many recent studies on PLP have investigated the relationship between cortical reorganization and PLP with the objective of discerning new ways to minimize pain in the residual limb in amputees. However, this approach has not been successful in describing the changes that occur in the peripheral or the central nervous systems and have not been able to concretely link any changes to PLP. Studying patients undergoing brachial plexus anesthesia (BPA) prior to upper extremity surgery has the potential to aid in the understanding of cortical remapping and the roles of the peripheral and central nervous systems in not only PLP but PLS as well. During upper extremity surgery, there have been reports that patients do not sense repositioning of the upper limb by the surgeon after BPA takes effect. This is similar to the phenomenon of the immobile, "frozen" limb occasionally experienced by major limb amputees. The purpose of this study is to investigate whether phantom limb pain and/or sensations can arise after induction of BPA prior to upper extremity surgery. In addition, this study aims to investigate if there is cortical remapping of the hand sensation onto the face before and after surgery. The outcome of this research will provide insight into the characteristics of cortical reorganization and how this correlates to phantom limbs, phantom pain, and hand-to-face remapping.
3. Study/Project Population, The general subject population includes male and female subjects greater than 18 years of age who are receiving BPA for the purposes of upper extremity surgery. Since this is a pilot study, we seek to recruit thirty (30) patients.
4. Research Design, To complete this study, a sensory map of participants' facial responses to the brushing of a Q-tip will be collected by a researcher before, and again after, BPA has been induced. In addition, follow-up phone sessions will be conducted on the day after surgery while BPA is still in effect, and daily, up to seven days, to identify whether participants are experiencing any changes in hand-to-face remapping should it be detected. This will be used to determine if cortical remapping has occurred as well as the time course of onset and reversal.
5. Study/Project Procedures, During the consent process all sections of the study will be described in detail. Participants will be able to determine if they can and would like to be enrolled in the study, Phantom Limb Experience After Brachial Plexus Anesthesia. 30 patients undergoing BPA in preparation for upper extremity surgery will be recruited for up to 10 data collection sessions. The first session will take place before the administration of BPA. The next sessions will occur after the administration of BPA and prior to surgery. A third session will occur after surgery is completed and prior to discharge home. Once the patient is discharged, follow-up phone sessions will be conducted in order to determine if hand-to-face remapping has occurred overnight and what the time course of onset and reversal of remapping and reorganization is. After obtaining informed consent, facial mapping of the patient's responses to light touch will be collected. To do this, a researcher will brush a Q-tip over all areas of the face, beginning at the forehead and working down towards the chin, while the participant's eyes are closed. During this process, the participant will be required to inform the researcher where the perception of brushing is being felt. During the follow-up phone sessions, the patient will answer questions about phantom limb sensations and pain, and will also be asked to touch different areas of his/her own face and report where the sensations are being perceived.
6. Outcome Measures. Data will be collected in the form of a verbal report. Participants will be instructed to inform researchers about the location that the brushing sensation is portrayed. In addition any feeling of phantom sensations or pain will also be recorded. Verbal reports will be collected at all in person sessions as well as phone follow us sessions. Analysis of these reports will include: the determination of the presence or absence of hand to face remapping, a detailed time course of onset and reversal if it occurs, specific locations of the hand-to-face remapping, changes in location of sensation reports prior to and following BPA, presence or absence of phantom limb sensations, such as the inability to feel limb repositioning, as well as the presence or absence of PLP. If PLP is experienced, scores of overall pain ratings will be conducted using a 10-cm visual analogue scale composed of a linear line where one end is labeled "no pain" and the other end is labeled "worst pain possible."

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects receiving brachial plexus anesthesia prior to upper extremity surgery
* Age 18 years or greater
* Ability to undergo 5-10 minutes of testing for multiple sessions: before anesthesia, following anesthesia but before surgery, following surgery while anesthesia remains effective, and throughout return of normal sensation
* Likely to complete all required sessions

Exclusion Criteria:

* Age less than 18 years old
* Physical or mental health condition which may interfere with being able to complete all required sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient already receiving BPA as a part of a previously planned shoulder surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-08-08 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Verbal Report | 3 days
  descriptions of sensations

SECONDARY OUTCOMES:
Visual analog scale | 3 days
  100mm line, no pain on one end, worst pain of life of another end. Participants mark spot on line. Answers are reported as a measure from the no pain end of the line.

CONTACTS AND LOCATIONS:
Locations (1):
- UTHSC, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided